CLINICAL TRIAL: NCT03104972
Title: Non-invasive Brain Stimulation for Pediatric ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Mor Nahum, Computerized Neurotherapy Lab, Hebrew University of Jerusalem
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HMO-17-0180
Record Dates: First submitted 2017-03-28; First posted 2017-04-07 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: ADHD
Keywords: ADHD; TRANS CRANIAL ELECTRIC STIMULATION
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: 'tDCS-tRNS' arm: a randomized controlled crossover study. 'tRNS-Sham' arm: a randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS - placebo (Experimental): tDCS-placebo (sham) group to receive either transcranial direct stimulation (tDCS) or matching placebo (sham( during 5 following days (one session each day). After a one week break, there will be a crossover between the control group and the sham group: those we received tDCS in the 1st week will get sham, while those who received sham in the 1st week will received tDCS at the 3rd week.
  Interventions: Device: tDCS; Device: sham
- tRNS - placebo (Experimental): trans cranial random stimulation (tRNS)-sham group, who will receive the same type of intervention with the same intervals as above but with tRNS instead of tDCS.
  Interventions: Device: tRNS; Device: sham
- tDCS-tRNS (Experimental): tDCS-tRNS group. Here the same intervention as above will be provided with the same intervals, but real tDCS and real tRNS will be provided in a counterbalanced fashion. This would allow to compare the different treatment in a within-subject design, as well as to compare the effect of those to sham stimulation in the first two groups in a between-subject design.
  Interventions: Device: tDCS; Device: tRNS

INTERVENTIONS:
Device: tDCS — Stimulation would be applied using semi-dry 5X5 cm electrodes. The current would be 0.75mA, which based on previous computational modeling of tDCS in children and is estimated to equal that of 1-1.5 mA in adults. This decision was made after considering the parameters that would influence current distribution and density at the site of stimulation such as thinner scalp, less cerebrospinal fluid, and smaller head size of the paediatric population. A similar dosage using tDCS was well tolerated by children, and was not associated with adverse effects29. The anodal electrode will be positioned above the dlPFC (F3 based on the International 10-20 system, while the cathodal electrode would be placed over the right supraorbital.
  Arms: tDCS - placebo; tDCS-tRNS
Device: tRNS — Children in the active tRNS group will received 0.75mA of tRNS (100-640Hz) to their left dorsolateral prefrontal cortex (dlPFC) and the right inferior frontal gyrus (IFG) via semi-dry 5cm X 5cm electrodes, attached under designated electrode positions (F3, F8) of a tES cap that followed the International 10-20 system (InnoSphere Inc., Haifa). The left dlPFC and right IFG were chosen, based on their contribution in executive control and inhibition. tRNS will be applied for 20 minutes per session during an iPad cognitive training. Similar duration has also been used in paediatrics using tDCS29. Similar to a previous tRNS study in children, and the rational provided for tDCS we will apply 0.75mA.
  Arms: tDCS-tRNS; tRNS - placebo
Device: sham — For sham-tRNS we will use the same montage as in active tRNS. For sham-tDCS we will use the same montage as in active tDCS. The only difference between active and sham tES would be that in the case of the sham tES the 30 sec of ramp up of the current from 0 to 0.75mA would not be followed by 19 min of stimulation at 0.75mA as in active tES, but would immediately be followed by 30 sec ramp down period to 0mA. Such method has been shown to provide effective blindness of the stimulation condition as both active and sham tES would lead to slight itching sensation that would disappear due scalp habitation. No further stimulation would be provided in the sham group during the daily session.
  Arms: tDCS - placebo; tRNS - placebo

SUMMARY:
The possibility of influencing brain activity and steadily enhancing behavioral performance through external intervention has long fascinated neuroscientists. One of these techniques, transcranial electrical stimulation (tES), has received great interest. Transcranial electrical stimulation (tES) in the current research includes two types of stimulation: transcranial direct current stimulation (tDCS) and transcranial random noise stimulation (tRNS).

The tES techniques involve the application of constant weak direct current (e.g. 1-2 mA) to the brain via skin-electrode interface, creating electric field that modulates neuronal activity. The safety profile of tES is excellent.

Despite effective pharmacotherapy for ADHD there is a need for improvement of cognitive dysfunction and behavioral symptoms that are only inadequately covered by pharmacological or psycho-social interventions. Since ADHD is the most common neurodevelopmental disorder in childhood with significant negative lifetime outcomes, non-invasive brain stimulation methods have been investigated in childhood and adolescents neuropsychiatric disorders showing promising results.

If tES is significantly effective for certain symptoms of ADHD, it may offer many advantages as a therapy. Treatment of ADHD with non-invasive brain stimulation has recently been reviewed in the medical literature, concluding that this technique seems to have efficacy in ADHD, however, standardized study protocols are needed to determine it.

In this study we intend to further examine the efficacy of tDCS and tRNS for children with ADHD and its effect on ADHD symptoms, memory, executive functions, in a randomized controlled crossover study.

DETAILED DESCRIPTION:
External influences on neuroplastic processes may be used for functional improvement of diseases, in particular for improving cortical functions. The possibility of influencing brain activity and steadily enhancing behavioral performance through external intervention has long fascinated neuroscientists. One of these techniques, transcranial electrical stimulation (tES), has received great interest because it has great potential use in basic research and clinical applications. Transcranial electrical stimulation (tES) in the current research includes two types of stimulation: transcranial direct current stimulation (tDCS) and transcranial random noise stimulation (tRNS). The tES techniques involve the application of constant weak direct current (e.g. 1-2 mA) to the brain via skin-electrode interface, creating electric field that modulates neuronal activity. This modulation is polarity dependent toward depolarization after anodal stimulation (excitatory) and toward hyperpolarization after cathodal stimulation (inhibitory), leading to transient changes in the resting membrane potential. The cumulative effect of longer stimulation results in a polarity-dependent facilitation or inhibition of the spontaneous neuronal firing rate and is considered neuromodulatory.

tDCS, provokes a sub-threshold modulation of neuronal excitability without depolarizing action potentials5. Post stimulation effects of tDCS depends on the duration of stimulation (lasting from several minutes up to hours) and can be found in the areas under the electrodes and also remote by network changes.

The mechanism by which tRNS influences brain activity differs from tDCS. The delivery of tRNS uses the same equipment as for tDCS. In tRNS, however, both electrodes can be used to stimulate either in homologous locations bilaterally or at different regions simultaneously. tRNS can be used to stimulate a region with a current that varies randomly in time. Such stimulation can induce excitability that lasts up to 60 minutes per 10 minutes of stimulation1. The most beneficial type of tRNS is at high-frequency (100-640Hz).

This is a randomized, double blinded, placebo-controlled, crossover study in ADHD children. Eligible participants will be randomized into the 3 following groups:

1. tDCS-placebo (sham) group to receive either tDCS or matching placebo (sham( during 5 following days (one session each day). After a one week break, there will be a crossover between the control group and the sham group: those we received tDCS in the 1st week will get sham, while those who received sham in the 1st week will received tDCS at the 3rd week.
2. tRNS-sham group, who will receive the same type of intervention with the same intervals as above but with tRNS instead of tDCS.
3. tDCS-tRNS group. Here the same intervention as above will be provided with the same intervals, but real tDCS and real tRNS will be provided in a counterbalanced fashion. This would allow to compare the different treatment in a within-subject design, as well as to compare the effect of those to sham stimulation in the first two groups in a between-subject design.

The total duration of subject participation will be 4 weeks. The study is conducted in the ADHD clinic of the Neuro-Cognitive Centre, at Hadassah-Hebrew University Medical Center.

tDCS: Stimulation would be applied using semi-dry 5X5 cm electrodes. The current would be 0.75mA, which based on previous computational modeling of tDCS in children and is estimated to equal that of 1-1.5 mA in adults. This decision was made after considering the parameters that would influence current distribution and density at the site of stimulation such as thinner scalp, less cerebrospinal fluid, and smaller head size of the paediatric population. A similar dosage using tDCS was well tolerated by children, and was not associated with adverse effects29. The anodal electrode will be positioned above the dlPFC (F3 based on the International 10-20 system, while the cathodal electrode would be placed over the right supraorbital. tRNS: Children in the active tRNS group will received 0.75mA of tRNS (100-640Hz) to their left dorsolateral prefrontal cortex (dlPFC) and the right inferior frontal gyrus (IFG) via semi-dry 5cm X 5cm electrodes, attached under designated electrode positions (F3, F8) of a tES cap that followed the International 10-20 system (InnoSphere Inc., Haifa). The left dlPFC and right IFG were chosen, based on their contribution in executive control and inhibition. tRNS will be applied for 20 minutes per session during an iPad cognitive training. Similar duration has also been used in paediatrics using tDCS29. Similar to a previous tRNS study in children, and the rational provided for tDCS we will apply 0.75mA.

Sham: For sham-tRNS we will use the same montage as in active tRNS. For sham-tDCS we will use the same montage as in active tDCS. The only difference between active and sham tES would be that in the case of the sham tES the 30 sec of ramp up of the current from 0 to 0.75mA would not be followed by 19 min of stimulation at 0.75mA as in active tES, but would immediately be followed by 30 sec ramp down period to 0mA. Such method has been shown to provide effective blindness of the stimulation condition as both active and sham tES would lead to slight itching sensation that would disappear due scalp habitation. No further stimulation would be provided in the sham group during the daily session.

The study will include 60 boys aged 7 to 12 years. The participants will be recruited among children referred to the clinic by pediatricians, general practitioners, teachers, psychologists or parents.

ELIGIBILITY:
Inclusion Criteria:

1. Meet ADHD criteria according to the DSM-5
2. Meet ADHD criteria according to "gold standard" AAP criteria = semi-structured interview, medical/neurological examination
3. Score above the standard clinical cut off values for ADHD symptoms on ADHD-RS
4. Drug naïve. -

Exclusion Criteria:

1. Chronic neurological disease
2. Epilepsy in subject or first degree relative
3. Intellectual disability
4. Any other chronic conditions
5. Chronic use of medications
6. Other primary psychiatric diagnosis (e.g., depression, anxiety, psychosis) -

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
ADHD Rating Scale (ADHD-RS) parameters | 4 weeks
  Assessment before and after intervention

SECONDARY OUTCOMES:
Wechsler Intelligence Scale for Children (WISC-IV) | 4 weeks
  All these parametres are part of the same scale (WISC-IV) including - Digit Span, Coding, Letter-Numbering Sequencing, Symbol Search. Assessment before and after intervention.
Behavior Rating Inventory of Executive Function (BRIEF) | 4 weeks
  Assessment before and after intervention
MOXO-Continuous Performance Test standardized attention test | 4 weeks
  Assessment before and after intervention

OTHER OUTCOMES:
Resting state Electroencephalography (EEG) | 4 weeks
  Assessment before and after intervention
CGI-S Scale = Clinical Global Impression - Severity | 4 weeks
  Assessment before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Computerized Neurotherapy Lab, School of OT, Hebrew University, Jerusalem, Mount Scopus, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berger I, Dakwar-Kawar O, Grossman ES, Nahum M, Cohen Kadosh R. Scaffolding the attention-deficit/hyperactivity disorder brain using transcranial direct current and random noise stimulation: A randomized controlled trial. Clin Neurophysiol. 2021 Mar;132(3):699-707. doi: 10.1016/j.clinph.2021.01.005. Epub 2021 Jan 27. PMID 33561725
- [Background] Dakwar-Kawar O, Berger I, Barzilay S, Grossman ES, Cohen Kadosh R, Nahum M. Examining the Effect of Transcranial Electrical Stimulation and Cognitive Training on Processing Speed in Pediatric Attention Deficit Hyperactivity Disorder: A Pilot Study. Front Hum Neurosci. 2022 Jul 27;16:791478. doi: 10.3389/fnhum.2022.791478. eCollection 2022. PMID 35966992
- Available data/document: similar protocol — http://www.ncbi.nlm.nih.gov/pubmed/27339019 — Looi CY, Cohen Kadosh R. Brain stimulation, mathematical, and numerical training: Contribution of core and noncore skills. Prog Brain Res. 2016;227:353-88. doi: 10.1016/bs.pbr.2016.04.009.